CLINICAL TRIAL: NCT05752357
Title: Does Circulating Tumor Cells Provide Diagnostic and Prognostic Roles in Peritoneal Carcinomatosis, Recurrence and Metastasis in Gastric Cancer, Pre-operatively and Postoperatively?
Brief Title: The Role of Pre-operative and Post-operative Circulating Tumor Cells in Gastric Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202100832B0
Record Dates: First submitted 2023-02-08; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma
Keywords: Circulating tumor cells; gastric cancer; peritoneal carcinomatosis; recurrence; metastasis
MeSH Terms: conditions — Carcinoma; Neoplastic Cells, Circulating; Stomach Neoplasms; Peritoneal Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm, observational arm: Patients who received surgery will routinely followed up by pre-op CTC, post-op CTC until 6 months after surgery.

SUMMARY:
In resectable gastric cancer participants who received curative surgery, to early and more accurately detect peritoneal carcinomatosis or occult metastasis is important. Also, investigators will look at CTC numbers in different timings after operation, to investigate the possibility of early detection for peritoneal carcinomatosis or occult metastasis. Also, this study will correlate the relationship of CTC and participants' survival.

DETAILED DESCRIPTION:
Circulating tumor cells (CTCs) are an emerging "liquid biopsy" that provide prognostic value for various types of solid cancer on early recurrence and survival. The evaluation of CTCs might be a useful strategy to predict tumor progression and prognosis in Gastric adenocarcinoma (GC). Previous study has shown that the frequency of CTC detection was higher in advanced GC than early GC, in poorly differentiated GC than well/moderately differentiated GC, and in GC with lymphatic metastasis than that without lymphatic metastasis. However, the impact of CTCs in the detection of PM in GC is still under debate. Peritoneal metastasis (PM) is highly related to recurrence and metastasis in GC; therefore, it was significantly related to disease free and overall survival of participants.

Consequently, several important questions and goals will be answered by this study:

To elucidate the clinical relationship between CTCs and PM in GCs before the operation; therefore, it could be an indicator of prophylactic during operation, which may possibly prolong the disease free and overall survival.

To establish a good model to follow-up a specific surface marker on CTCs, which could be possibly utilized as a more sensitive marker, comparing with CEA or image study, to more accurately detect the early recurrence or metastasis in GC.

To verify that dynamically monitoring CTCs status and changes during long-term follow-up and anti-cancer treatment are feasible and clinically meaningful to survival or treatment responses.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling 150 cases
* Stage I or more advanced gastric cancer, pathology proved
* Diagnosed at age ≥ 20 years
* Enrolled before surgery at the General Surgery Department, both inpatient and outpatient services.

Exclusion Criteria:

* Patient's refusal
* Poor compliance, unable to cooperate for blood sampling for CTC isolation as time schedule or clinical treatment or follow-up
* Difficult blood sampling
* No more needs for CTCs evaluation, decided by clinicians.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In resectable gastric cancer patients, who undergo radical intent gastrectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of disease recurrence | Baseline
  Circulating tumor cells detection in different time after operation, to evaluate the clinical relationship between Circulating tumor cells and disease recurrence.
Percentage of disease recurrence | Post-operation within 3 days
  Circulating tumor cells detection in different time after operation, to evaluate the clinical relationship between Circulating tumor cells and disease recurrence.
Percentage of disease recurrence | Post-operation day 4 - 4 weeks
  Circulating tumor cells detection in different time after operation, to evaluate the clinical relationship between Circulating tumor cells and disease recurrence.
Percentage of disease recurrence | Post-operation 3 months
  Circulating tumor cells detection in different time after operation, to evaluate the clinical relationship between Circulating tumor cells and disease recurrence.
Percentage of disease recurrence | Post-operation 6 months
  Circulating tumor cells detection in different time after operation, to evaluate the clinical relationship between Circulating tumor cells and disease recurrence.

SECONDARY OUTCOMES:
Percentage of peritoneal seedings | Baseline
  Circulating tumor cells detection in different time after operation, to early detect peritoneal carcinomatosis or occult metastasis.
Percentage of peritoneal seedings | Post-operation within 3 days
  Circulating tumor cells detection in different time after operation, to early detect peritoneal carcinomatosis or occult metastasis.
Percentage of peritoneal seedings | Post-operation day 4 - 4 weeks
  Circulating tumor cells detection in different time after operation, to early detect peritoneal carcinomatosis or occult metastasis.
Percentage of peritoneal seedings | Post-operation 3 months
  Circulating tumor cells detection in different time after operation, to early detect peritoneal carcinomatosis or occult metastasis.
Percentage of peritoneal seedings | Post-operation 6 months
  Circulating tumor cells detection in different time after operation, to early detect peritoneal carcinomatosis or occult metastasis.
overall survival time | Post-operation 1 year.
  To correlate the relationship of circulating tumor cells and long-term survival time.
overall survival time | Post-operation 2 year.
  To correlate the relationship of circulating tumor cells and long-term survival time.
Progression-free survival | Post-operation 1 year.
  To correlate the relationship of circulating tumor cells and Progression-free survival.
Progression-free survival | Post-operation 2 year.
  To correlate the relationship of circulating tumor cells and Progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chun Chang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan